CLINICAL TRIAL: NCT00642850
Title: A Single Arm, Open Label Study to Assess the Efficacy, Safety and Tolerability of Once-monthly Administration of Intravenous C.E.R.A. for the Maintenance of Haemoglobin Levels in Dialysis Patients With Chronic Renal Anaemia
Brief Title: STABIL Study: National Study With Mircera for Maintenance of Hemoglobin Level in Dialysis Patients
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ML21040
Record Dates: First submitted 2008-03-19; First posted 2008-03-25 (Estimated); Results first posted 2016-06-23 (Estimated); Last update posted 2016-06-23 (Estimated); Status verified 2016-05

CONDITIONS: Anemia
MeSH Terms: conditions — Anemia | interventions — continuous erythropoietin receptor activator

ARMS (1):
- 1 (Experimental)
  Interventions: Drug: methoxy polyethylene glycol-epoetin beta [Mircera]

INTERVENTIONS:
Drug: methoxy polyethylene glycol-epoetin beta [Mircera] — 120, 200 or 360 micrograms iv monthly (starting dose)

SUMMARY:
This single arm study will assess the efficacy, safety and tolerability of once-monthly administration of intravenous Mircera for the maintenance of hemoglobin levels in dialysis participants with chronic renal anemia. Participants will receive monthly intravenous injections of Mircera, at a starting dose of 120, 200 or 360 micrograms, according to the dose of epoetin administered in the week preceding first study drug administration. The anticipated time on study treatment is 3-12 months, and the target sample size is 100-500 individuals.

ELIGIBILITY:
Inclusion Criteria:

* Chronic renal anemia;
* Continuous stable intravenous maintenance epoetin therapy during previous month;
* Regular long-term hemodialysis therapy with the same mode of dialysis for previous 3 months.

Exclusion Criteria:

* Transfusion of red blood cells during previous 2 months;
* Poorly controlled hypertension, that is, sitting blood pressure exceeding 170/100 millimeter of mercury (mmHg) despite medication;
* Significant acute or chronic bleeding.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 188 (Actual)
Dates: Start 2007-11; Primary Completion 2009-07 (Actual); Study Completion 2009-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (21):
- Czechia (21):
  - Brno
  - Český Krumlov
  - Děčín
  - Havířov
  - Hradec Králové
  - Jihlava
  - Karlovy Vary
  - Kolin III
  - Liberec
  - Nový Jičín
  - Olomouc
  - Ostrava
  - Písek
  - Prague
  - Strakonice
  - Šumperk
  - Tábor
  - Teplice
  - Třebíč
  - Ústí nad Labem
  - Znojmo

REFERENCES:
- [Derived] Locatelli F, Choukroun G, Truman M, Wiggenhauser A, Fliser D. Once-Monthly Continuous Erythropoietin Receptor Activator (C.E.R.A.) in Patients with Hemodialysis-Dependent Chronic Kidney Disease: Pooled Data from Phase III Trials. Adv Ther. 2016 Apr;33(4):610-25. doi: 10.1007/s12325-016-0309-6. Epub 2016 Mar 10. PMID 26965694

RESULTS

PARTICIPANT FLOW:
Groups:
- C.E.R.A.: Adult participants with chronic renal disease and who had received intravenous epoetin (epoetin alfa, epoetin beta or darbepoetin alfa) maintenance treatment, received (after fulfilling all inclusion/exclusion criteria and 4 weeks stability verification period) intravenous methoxy polyethylene glycol-epoetin beta (C.E.R.A.) at starting dose of 120, 200, or 360 microgram (mcg) every 4 weeks for 24 weeks.
Period: Overall Study
Arm/Group | C.E.R.A.
Started | 188
Completed | 155
Not Completed | 33
Not completed — Death | 7
Not completed — Adverse Event | 2
Not completed — Lack of Efficacy | 1
Not completed — Protocol Violation | 2
Not completed — Kidney transplantation | 8
Not completed — Blood transfusion | 6
Not completed — Other reasons | 7

BASELINE CHARACTERISTICS:
Population: The safety population was defined as all participants enrolled into the study.
Groups:
- C.E.R.A.: Adult participants with chronic renal disease and who had received intravenous epoetin maintenance treatment, received intravenous C.E.R.A. at starting dose of 120, 200, or 360 mcg every 4 weeks for 24 weeks.
Arm/Group | C.E.R.A.
Number analyzed (Participants) | 188
Age, Continuous [Mean (Standard Deviation); unit: years] | 64.9 (11.56)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 84
  Male | 104

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants Maintaining Average Hemoglobin Concentration Within +/-1 Gram Per Deciliter (g/dL) of Reference and Within the Target Range
Description: Percentage of participants maintaining their mean hemoglobin concentration in g/dL within plus or minus (+/-) 1 g/dL of their reference hemoglobin value, and between the target range of 10.0 and 12.0 g/dL during the efficacy evaluation period (EEP). The reference hemoglobin value was defined on the basis of the 5 assessments recorded during the Stability Verification Period (SVP) at Weeks -4, -3, -2, -1 and 0. The mean hemoglobin concentration for each individual participant during the EEP (Week 17 up to Week 24) was estimated as a time adjusted average.
Time Frame: Week 17 up to Week 24
Population: Per protocol (PP) population included all participants in the safety population with the exception of participants with less than 3 recorded hemoglobin values, missing administrations of C.E.R.A., withdrawal, inadequate iron status in Weeks 16-24.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | C.E.R.A.
Number analyzed (Participants) | 154
percentage of participants | 53.3 [45.1 to 61.3]

2. Secondary Outcome: Change in Hemoglobin Concentration Between Reference (SVP) and EEP
Description: The mean change of the time adjusted average of hemoglobin from reference value obtained during the SVP (Week -4 up to Week -1) and the value during EEP (Week 17 up to Week 24) was assessed.
Time Frame: Week -4 up to Week -1 and Week 17 up to Week 24
Population: The Intention-to-treat (ITT) population included all participants who had received at least 1 dose of C.E.R.A. (Week 0) and for whom data for at least 1 follow-up variable had been available.
Measure: Mean (Standard Deviation); unit: g/dL
Arm/Group | C.E.R.A.
Number analyzed (Participants) | 186
g/dL | 0.0 (1.21)

3. Secondary Outcome: Percentage of Participants Maintaining Hemoglobin Concentration Within the Target Range During EEP
Description: Percentage of participants maintaining hemoglobin concentration within the target range of 10.0 to 12.0 g/dL during EEP (Week 17 to Week 24) was assessed.
Time Frame: Week 17 up to Week 24
Population: ITT Population.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | C.E.R.A.
Number analyzed (Participants) | 186
percentage of participants | 57.0 [49.5 to 64.2]

4. Secondary Outcome: Mean Time Spent by Participants With Hemoglobin Concentration in the Target Range During the EEP
Description: Mean time spent by participants with hemoglobin concentration in the target range of 10.0 to 12.0 g/dL during the EEP (Week 17 to Week 24) was assessed.
Time Frame: Week 17 up to Week 24
Population: ITT Population.
Measure: Mean (Standard Deviation); unit: days
Arm/Group | C.E.R.A.
Number analyzed (Participants) | 186
days | 32 (18.4)

5. Secondary Outcome: Percentage of Participants Requiring Any Dose Adjustment
Description: Percentage of participants requiring adjustment in the dose of study drug during the dose titration period (DTP: Week 1 to Week 16) and EEP (Week 17 to Week 24) was reported.
Time Frame: Week 1 to Week 16 and Week 17 to Week 24
Population: ITT Population. Here, 'N' (number of participants analyzed) signifies the number of participants evaluable for this outcome measure and 'n' signifies the number of participants evaluable for specified category.
Measure: Number; unit: percentage of participants
Arm/Group | C.E.R.A.
Number analyzed (Participants) | 186
percentage of participants
  DTP (n = 186) | 75.0
  EEP (n = 165) | 32.0

6. Secondary Outcome: Number of Participants With Red Blood Cell Transfusion During the Study
Description: Number of participant who underwent red blood cell transfusion during the study was reported.
Time Frame: Week -4 up to Week 28
Population: ITT Population.
Measure: Number; unit: participants
Arm/Group | C.E.R.A.
Number analyzed (Participants) | 186
participants | 9

7. Secondary Outcome: Number of Participants With Anti-epoetin Antibody
Time Frame: Week -4 and at early withdrawal or Week 28
Population: ITT Population.
Measure: Number; unit: participants
Arm/Group | C.E.R.A.
Number analyzed (Participants) | 186
participants
  Week -4 | 0
  Early Withdrawal or Week 28 | 0

ADVERSE EVENTS:
Time Frame: Up to 28 weeks
Description: Only adverse events with an onset date after the start of medication included.
Arm/Group | C.E.R.A.
Serious Adverse Events (participants affected / at risk) | 41/188
Other Adverse Events (participants affected / at risk) | 38/188
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | C.E.R.A. (N=188)
Angina pectoris (Cardiac disorders) | 1
Atrial fibrillation (Cardiac disorders) | 2
Atrioventricular block (Cardiac disorders) | 1
Cardiac arrest (Cardiac disorders) | 1
Cardiac failure (Cardiac disorders) | 1
Myocardial ischaemia (Cardiac disorders) | 1
Ventricular fibrillation (Cardiac disorders) | 1
Coeliac artery stenosis (Gastrointestinal disorders) | 1
Dyspepsia (Gastrointestinal disorders) | 2
Gastric ulcer haemorrhage (Gastrointestinal disorders) | 1
Gastric ulcer perforation (Gastrointestinal disorders) | 1
Haemorrhoidal haemorrhage (Gastrointestinal disorders) | 1
Intestinal angina (Gastrointestinal disorders) | 1
Intestinal haemorrhage (Gastrointestinal disorders) | 1
Sudden death (General disorders) | 1
Arteriovenous fistula site infection (Infections and infestations) | 1
Bronchitis (Infections and infestations) | 2
Catheter sepsis (Infections and infestations) | 2
Chlamydial infection (Infections and infestations) | 1
Gastroenteritis (Infections and infestations) | 1
Haematoma infection (Infections and infestations) | 1
Herpes zoster (Infections and infestations) | 1
Sepsis (Infections and infestations) | 2
Wound infection staphylococcal (Infections and infestations) | 1
Accident (Injury, poisoning and procedural complications) | 1
Arteriovenous fistula site complication (Injury, poisoning and procedural complications) | 1
Complications of transplanted kidney (Injury, poisoning and procedural complications) | 1
Concussion (Injury, poisoning and procedural complications) | 1
Femur fracture (Injury, poisoning and procedural complications) | 1
Graft complication (Injury, poisoning and procedural complications) | 1
Humerus fracture (Injury, poisoning and procedural complications) | 1
Post procedural haemorrhage (Injury, poisoning and procedural complications) | 1
Arteriogram (Investigations) | 1
Arteriogram coronary (Investigations) | 2
Fluid retention (Metabolism and nutrition disorders) | 1
Polymyalgia rheumatica (Musculoskeletal and connective tissue disorders) | 1
Spondylolisthesis (Musculoskeletal and connective tissue disorders) | 1
Benign pancreatic neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Lung carcinoma cell type unspecified stage III (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Carotid artery stenosis (Nervous system disorders) | 1
Cerebral haemorrhage (Nervous system disorders) | 2
Cerebrovascular accident (Nervous system disorders) | 1
Subarachnoid haemorrhage (Nervous system disorders) | 1
Transient ischaemic attack (Nervous system disorders) | 1
Breast dysplasia (Reproductive system and breast disorders) | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1
Hydrothorax (Respiratory, thoracic and mediastinal disorders) | 2
Dry gangrene (Skin and subcutaneous tissue disorders) | 1
Arteriovenous fistula operation (Surgical and medical procedures) | 1
Coronary artery bypass (Surgical and medical procedures) | 1
Surgery (Surgical and medical procedures) | 1
Aneurysm ruptured (Vascular disorders) | 1
Hypertension (Vascular disorders) | 1
Shock (Vascular disorders) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | C.E.R.A. (N=188)
Diarrhoea (Gastrointestinal disorders) | 11
Bronchitis (Infections and infestations) | 10
Hypertension (Vascular disorders) | 22

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Study being conducted under this Agreement is part of the Overall Study. Investigator is free to publish in reputable journals or to present at professional conferences the results of the Study, but only after the first publication or presentation that involves the Overall Study. The Sponsor may request that Confidential Information be deleted and/or the publication be postponed in order to protect the Sponsor's intellectual property rights.